CLINICAL TRIAL: NCT01717794
Title: Prospective Randomized Trial on Total Laparoscopic Hysterectomy With Pelvic Lymphadenectomy for the Treatment of Endometrial Cancer FIGO Stage IB-II: Thunderbeat Technology Versus Standard Bipolar Electro-surgery.
Brief Title: Thunderbeat Technology vs Standard Bipolar Electro-surgery in Total Laparoscopic Hysterectomy With Pelvic Lymphadenectomy for Endometrial Cancer
Acronym: Thunder Endom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Director, Dip per la Tutela della Salute della Donna e della Vita Nascente, del Bambino e dell'Adolescente - Policlinico Gemelli, Rome, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Thunder Endometrium
Record Dates: First submitted 2012-10-28; First posted 2012-10-30 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Endometrial Cancer
Keywords: operative time; laparoscopy; total hysterectomy; pelvic lymphadenectomy; endometrial cancer; Thunderbeat
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard bipolar electrosurgery (Active Comparator): Laparoscopic total hysterectomy with pelvic lymphadenectomy are performed with standard bipolar electrosurgery.
  A 10 mm port is inserted at the umbilicus for the telescope. Once pneumoperitoneum (12 mmHg) is achieved, intra-abdominal visualization will be obtained with a 0° high-definition telescope.
  Two additional 5 mm ports are placed under direct visualization. One more 5-mm trocar is inserted in the right mid abdomen at the level of the umbilicus. The instruments used include bipolar grasper, monopolar scissors, monopolar hook, various graspers and a suction irrigation system.
  Interventions: Procedure: Standard bipolar electrosurgery
- Thunderbeat technology (Experimental): Laparoscopic total hysterectomy with pelvic lymphadenectomy are performed with Thunderbeat technology: using Thunderbeat technique, surgeons can avoid changing instruments during surgery since Thunderbeat combines bipolar energy for haemostasis and ultrasound for dissection and cut.
  Thunderbeat is used to coagulate the fallopian tubes, to coagulate and divide the round ligaments, to seal ovarian pedicles, to open the anterior and posteriors leaves of the broad ligaments peritoneum, to develop the paravesical and pararectal spaces, to seal uterine arteries and uterine pedicles, to incise the bladder peritoneum, to dissect the bladder, to develop rectovaginal septum, to cut parametria, and to divide the uterosacral ligaments. Thunderbeat is also used to perform the pelvic lymphadenectomy and, if necessary, the para-aortic lymphadenectomy.
  Interventions: Procedure: Thunderbeat technology

INTERVENTIONS:
Procedure: Thunderbeat technology
  Arms: Thunderbeat technology
Procedure: Standard bipolar electrosurgery
  Arms: Standard bipolar electrosurgery

SUMMARY:
This prospective randomized pilot study is aimed to verify if the operative time of a TLH with pelvic lymphadenectomy for endometrial cancer FIGO stage IB-II could be reduced using Thunderbeat (an ultrasonic energy device that incises and coagulates by using ultrasonic and bipolar technology ) (Olympus Medical Systems Corp, Tokyo) vs. bipolar electrosurgery .

Secondary endpoints of this comparison are incidence of intra- or postoperative complications (Cardiac, Respiratory, Neurological, Gastrointestinal, Renal, Fever, Wound or other Infection, Lymphocele), estimated blood loss, postoperative pain (evaluated by VAS), days of hospitalization and costs for the health care system.

DETAILED DESCRIPTION:
The standard treatment for early-stage endometrial cancer is surgery. Surgical procedures include washing for cytology, total extrafascial hysterectomy and bilateral salpingo-oophorectomy. Although the therapeutic value of routine pelvic and para-aortic lymphadenectomy is debated, staging information is a critical determinant of adjuvant therapy for most gynecologic oncologists.

Type-1 endometrial cancer spread is limited to the pelvic nodes in most cases. If there are positive lymph nodes, those around the obturator nerve and around the external and common iliac vessels are more likely to be involved than those in the presacral area. Isolated involvement of the para-aortic nodes is rare. Complete excision of the nodes located around the iliac vessels and above the obturator nerve allows identiﬁcation of 90% of node-positive patients.

The decision on whether to undertake lymphadenectomy should not be based on palpation of the nodal area, because less than 10% of patients with nodal metastases have grossly enlarged nodes.

Patients with endometrioid cancer, grade 1-2 with deep myometrial invasion and any grade 3 endometrioid endometrial cancer have at least a 5% risk of having positive pelvic lymph nodes. In our current treatment protocol, these patients undergo complete pelvic lymphadenectomy. Laparotomy may be indicated in endometrial cancer patients presenting with grossly positive pelvic nodes, grossly positive adnexal metastasis, or serosal inﬁltration.

Although the complication rate of a simple hysterectomy with bilateral salpingo-oophorectomy is not very high, over 70% new cases of endometrial cancer are diagnosed in post-menopausal women, commonly associated with medical co-morbidities, such as diabetes, hypertension and obesity. Abdominal surgery therefore exposes them to an increased risk of complications. Vaginal hysterectomy has been suggested as an attractive alternative to abdominal surgery for these patients, but this approach does not allow exploration of the abdominal cavity, peritoneal washing, and lymph-node dissection. Laparoscopic-assisted vaginal hysterectomy or total laparoscopic hysterectomy overcome the previous limitations.

In 1993, Childers et al first proposed laparoscopy as an option for early-stage endometrial cancer. Despite its recognized benefits, many surgeons found this approach difficult for routine use such that relatively few centers offered laparoscopic hysterectomy and lymphadenectomy for a majority of their patients.

From those first reports there have been 12 major reports on the use of laparoscopy, often comparing to series of similar patients staged by laparotomy. Clear advantages, such as the reduction of peri-operative complications, the shorter hospital stay and the earlier recovery, have been confirmed in each series. Failure to complete the staging procedure by laparoscopy ranges between 5 and 35% of the patients, most frequently due to obesity of the patients. In reality in 2005 some researchers have suggested that laparoscopic surgery is safe in obese or elderly patients with endometrial cancer too.

Moreover, this approach does not seem to modify the incidence of recurrence and overall patient survival. The big randomized trials planned to study differences in morbidity and survival between laparoscopy or laparotomy in endometrial cancer are the GOG LAP-2 study, the Dutch study from Bijen and Mourits, and the Australian study LACE. Unfortunately none of these three randomised trials have yet reported survival data, but only on health-related issues and complications. In the GOG study 33, patients with clinical stage I to IIA uterine cancer were randomly assigned to laparoscopy (n = 1,696) or open laparotomy (n = 920), including hysterectomy, salpingo-oophorectomy, pelvic cytology, and pelvic and para-aortic lymphadenectomy. Laparoscopy resulted in fewer postoperative moderate or severe adverse events, a shorter hospital stay, and a longer operative time than did laparotomy. The median operative time for the open laparotomy arm was 130 minutes (range 102-167 minutes), and for the laparoscopy arm, it was 204 minutes (rang 160-252 minutes; P < .001).

In the Dutch 34-35 study the major and minor complication rates were the same in the group of patients treated with laparoscopy compared with laparotomy. However, TLH was associated with less blood loss, less use of pain medication, a shorter hospital stay, and a longer operative time than with TAH. The median duration of surgery was 115 minutes in the TLH group, (range 35-267) and 71 minutes (range 31-239) in the TAH group. The difference with the GOG study is probably due to the fact that the patients in the Netherlands only underwent a hysterectomy and bilateral salpingo-oophorectomy and not a complete surgical staging including pelvic and para-aortic lymphadenectomy.

In the Australian LACE study 36 patients with stage I endometrioid adenocarcinoma were randomly assigned to TLH (n=190) or TAH (n=142). Surgeons were required to perform pelvic node (with or without) para-aortic lymph-node dissection as part of the treatment in both groups. Operating time was significantly longer in the TLH group (138 minutes [SD 43]) than in the TAH group (109 minutes [34]; p=0•001).

Health-related outcome was reported in all three trials. Better physical functioning, body image, reduced pain, and an earlier resumption of work over the 6-week post-laparoscopy period was reported in the GOG and the Dutch study than in the laparotomy patients, but these differences disappeared 6 months after surgery. In the Australian study, quality of life was still improved 6 months after surgery.

In conclusion, laparoscopic treatment of endometrial cancer clinically confined to the uterus is associated with less pain, shorter hospital stay, faster recovery, and better quality of life at least 3 months post surgery, but with a longer operative time than with laparotomy.

Another recent single institution Italian trial randomized patients with clinical stage I endometrial cancer to receive TLH (n=81) or TAH (n=78) with bilateral salpingo-oophorectomy and bilateral pelvic lymphadenectomy. 37 Para-aortic lymphadenectomy was performed in selected cases. The mean operative time was 123 minutes ± 29 (95% CI 111-198) in the LPT group and 136 minutes ± 31 (95% CI 118- 181) in the LPS group (P<0.01). These operative times match closely with our experience by both laparotomy and laparoscopy, using conventional bipolar electrosurgery.

Shortening the operative time of laparoscopy could further increase the benefits of the laparoscopic approach, especially in obese patients. Overweight (defined as body-mass index [BMI] of at least 25 kg/m2) is an important risk factor present in almost 50% of women with endometrial cancer.

Since these patients are characterised by several systemic physiopathological alterations, the perioperative management may present some problems, mainly related to their respiratory system (obstructive sleep apnea, airway intubation and atelectasis). Obstructive sleep apnea-hypopnea syndrome (OSA) occurs in up to 70% of morbidly obese patients undergoing surgery 39 being OSA a known risk factor for adverse perioperative outcomes.

Shortening the operative time could reduce these perioperative complications and the postoperative pain. This could translate in fewer days of hospitalization and than lower incidence of hospital infections and lower costs for the health care system.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Age ≤ 75 years
* Patient's informed consent
* American Society of Anesthesiologists: < class III or IV
* No actual pregnancies or P.I.D.
* No previous major abdominal surgical procedures
* Endometrial cancer FIGO stages IB-II
* Endometrioid histotype
* No previous radiotherapy on pelvic fields
* No uterine size larger than conform 10 weeks gestation

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Operative time for total laparoscopic hysterectomy with pelvic lymphadenectomy | 24 months
  Operative time will be calculated from the entrance in the abdominal cavity to the closure of the skin trocar accesses.

SECONDARY OUTCOMES:
Intra- or post operative complications | 24 months
  Cardiac, Respiratory, Neurological, Gastrointestinal, Renal, Fever, Wound or other Infection, Lymphocele

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred the Hearth, Rome, Italy